CLINICAL TRIAL: NCT07285460
Title: An Open-label, Parallel, Phase 3, Two-arm Study to Investigate the Efficacy and Safety of Fitusiran Prophylaxis in Male Participants Aged 1 to Less Than 12 Years With Hemophilia A or B With or Without Inhibitory Antibodies to Factors VIII or IX
Brief Title: A Study to Investigate the Efficacy and Safety of Fitusiran Prophylaxis in Male Participants Aged 1 to Less Than 12 Years With Hemophilia A or B
Acronym: ATLAS-KIDS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC17905; U1111-1280-7028 (Registry Identifier: ICTRP); 2025-521858-42 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-12-09; First posted 2025-12-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — fitusiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fitusiran-naïve arm (Experimental): Participants will go through a 24-week standard of care (SOC) period before receiving a selected dose of fitusiran at regular interval.
  If a fitusiran dose adjustment is needed during the study, participants will follow a specific dosing regimen as per study protocol.
  Interventions: Drug: Fitusiran; Biological: Clotting factor concentrates (CFC) or bypassing agents (BPA); Biological: Antithrombin concentrate (ATIIIC)
- EFC15647 roll-over arm (Experimental): Participants will continue receiving their current fitusiran dose from EFC15467.
  If a fitusiran dose adjustment is needed during the study, participants will follow a specific dosing regimen as per study protocol.
  Interventions: Drug: Fitusiran; Biological: Clotting factor concentrates (CFC) or bypassing agents (BPA); Biological: Antithrombin concentrate (ATIIIC)

INTERVENTIONS:
Drug: Fitusiran — Pharmaceutical form: solution for injection in PBS Route of administration: subcutaneous
  Other Names: SAR439774; Qfitlia™
Biological: Clotting factor concentrates (CFC) or bypassing agents (BPA) — Pharmaceutical form: solution for injection Route of administration: intravenous injection
Biological: Antithrombin concentrate (ATIIIC) — Pharmaceutical form: solution for injection Route of administration: intravenous injection

SUMMARY:
This is a parallel, Phase 3, two-arm, open-label study to evaluate the efficacy and safety of treatment with fitusiran prophylaxis administered to male pediatric participants (aged 1 to <12 years) who have severe hemophilia A or B, with or without inhibitory antibodies to FVIII or FIX.

Number of participants:

Approximately 85 participants will be enrolled into the study:

* Approximately 60 fitusiran-naïve participants with severe hemophilia A or B, with or without inhibitors (fitusiran-naïve arm), and
* Approximately 25 participants with severe hemophilia A or B with inhibitors rolling over from the EFC15467* dose confirmation study (roll-over arm).

  * Fitusiran has been investigated in the pediatric population in study EFC15467, which enrolled male participants aged 1 to <12 years with hemophilia A or B with inhibitors to examine the safety and tolerability of fitusiran in the pediatric population.

Participants will be enrolled into 1 of 2 arms:

* Fitusiran-naïve: these participants have not previously received fitusiran, and they will undergo screening and study eligibility assessments. Once enrolled, they will go through a 24-week standard of care (SOC) period before starting fitusiran prophylaxis.
* Roll-over participants from the EFC15467 study: only participants who are still on active treatment in study EFC15467 and consenting to study EFC17905 will be eligible to roll over. They will not need to undergo screening or further eligibility assessments. They will directly enroll into the fitusiran treatment period and continue treatment on their current fitusiran dose.

The duration of fitusiran treatment will be up to 160 weeks for the fitusiran-naïve arm and up to 60 weeks for the roll-over arm.

DETAILED DESCRIPTION:
The duration of fitusiran treatment will be up to 160 weeks for the fitusiran-naïve arm and up to 60 weeks for the roll-over arm.

ELIGIBILITY:
Inclusion Criteria:

Participants not previously exposed to fitusiran are eligible to be included in the study only if all of the following criteria apply:

* Participant must be 1 to <12 years of age at the time of enrollment.
* Participants must have severe hemophilia A or B (FVIII <1% or FIX ≤2%) as evidenced by a central laboratory measurement at screening or documented medical record evidence.
* Participants must meet inhibitor or non-inhibitor status as defined below:

Inhibitor:

Requiring use of BPA for prophylaxis or BPA as on-demand therapy for any bleeding episodes for at least the last 3 months prior to screening, and meet one of the following Nijmegen-modified Bethesda assay results criteria:

* Inhibitor titer of ≥0.6 BU/mL at screening, OR
* Inhibitor titer of <0.6 BU/mL at screening with medical record evidence of 2 consecutive titers ≥0.6 BU/mL, OR
* Inhibitor titer of <0.6 BU/mL at screening with medical record evidence of 1 inhibitor titer ≥0.6 BU/mL and a history of anamnestic response, or severe allergic reaction (eg, anaphylaxis) or nephrotic syndrome

Non-inhibitor:

Requiring use of clotting factor concentrates (CFCs) for prophylaxis or CFCs as on-demand therapy for any bleeding episodes for at least the last 3 months prior to screening, and meet each of the following criterion:

* Nijmegen-modified Bethesda assay inhibitor titer of <0.6 BU/mL at screening, AND
* No use of BPA to treat bleeding episodes for at least the last 3 months prior to screening

  * Participants must have adequate peripheral venous access, as determined by the Investigator, to allow the blood draws required by the study protocol.
  * Male: There are no contraceptive requirements for this study except where required by local regulations.
  * Capable of giving signed informed consent/assent. A signed written informed consent must be obtained from parent(s)/legal guardian (hereafter referred to as the "parent"), as well as a written or oral assent obtained from participant, per local and national requirements.

Exclusion Criteria:

Participants not previously exposed to fitusiran are excluded from the study if any of the following criteria apply:

* Known co-existing bleeding disorders other than hemophilia A or B.
* Presence of clinically significant liver disease.
* History of antiphospholipid antibody syndrome.
* History of arterial or venous thromboembolism, unrelated to an indwelling venous access
* Any condition (eg, medical concern), which in the opinion of the Investigator, would make the participant unsuitable for dosing or which could interfere with the study compliance, the participant's safety and/or the participant's participation in the completion of the treatment period of the study.
* History of multiple drug allergies or history of allergic reaction to an oligonucleotide or GalNAc.
* Subjects with a central or peripheral indwelling catheter, with a history of venous access complications (such as infections, thrombosis) leading to hospitalization and/or systemic anticoagulation therapy in the last 12 months.
* At screening, anticipated need of surgery during the study or planned surgery scheduled to occur during the study.
* Completion of a surgical procedure within 14 days prior to screening, or currently receiving additional BPA infusion for postoperative hemostasis.
* History of intolerance to SC injection(s).
* Current participation in ITI therapy.
* The use of emicizumab (Hemlibra®) or any non-factor bleed management treatment within 6 months prior to screening
* Prior gene therapy
* Current or future participation in another clinical study, scheduled to occur during this study, involving an investigational product other than fitusiran or an investigational device.
* AT activity <60% at screening, as determined by central laboratory analysis.
* Co-existing thrombophilic disorder.
* Presence of an active Hepatitis C virus infection
* Presence of acute hepatitis A or Hepatitis E virus infection.
* Presence of acute or chronic hepatitis B virus infection.
* Platelet count ≤100 000/μL.
* Presence of acute infection at screening.
* Human immunodeficiency virus (HIV) positive with a CD4 count of <400 cells/μL.
* Estimated glomerular filtration rate ≤45 mL/min/1.73 m2 (using the Schwartz formula).

Ages: 1 Year to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2029-08-04 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Annualized treated bleeding rate (ABR) in the fitusiran primary efficacy period and in the SOC period | Day 85 to Day 421 (fitusiran primary efficacy period); Day -168 to Day -1 (SOC period)
  A bleeding episode is defined as any occurrence of hemorrhage that requires administration of CFCs or BPAs

SECONDARY OUTCOMES:
Annualized spontaneous bleeding rate (AsBR) in the fitusiran primary efficacy period and in the SOC period | Day 85 to Day 421 (fitusiran primary efficacy period); Day -168 to Day -1 (SOC period)
  A spontaneous bleeding episode is a bleeding event that occurs for no apparent or known reason, particularly into the joints, muscles, and soft tissues
Annualized joint bleeding rate (AjBR) in the fitusiran primary efficacy period and in the SOC period | Day 85 to Day 421 (fitusiran primary efficacy period); Day -168 to Day -1 (SOC period)
  A joint bleeding episode is characterized by an unusual sensation in the joint ("aura") in combination with 1) increasing swelling or warmth over the skin over the joint, 2) increasing pain, or 3) progressive loss of range of motion or difficulty in using the limb as compared with baseline
ABR in the fitusiran treatment period (160 weeks) for fitusiran-naïve participants | Day 1 to Day 1121
  A bleeding episode is defined as any occurrence of hemorrhage that requires administration of CFCs or BPAs
ABR in the fitusiran treatment period (60 weeks) for rolled-over participants | Day 1 to Day 421
  A bleeding episode is defined as any occurrence of hemorrhage that requires administration of CFCs or BPAs
Change in physical activity | From Day 1 to Day 421; From Week -24 to Day -1
  Change in physical activity as measured via the PROMIS questionnaire
Change in pain intensity | From Day 1 to Day 421; From Week -24 to Day -1
  Change in pain intensity as measured via the PROMIS questionnaire
Change in HRQoL | From Day 1 to Day 421; From Week -24 to Day -1
  Change in HRQoL as measured by the EuroQoL 5-dimension questionnaire
Incidence, severity, seriousness, and relatedness of adverse events (AEs) | Date of signed ICF (Day -228 to Day -169) until last AT follow-up visit (Day 1121 + approximately 24 weeks)
  All AEs are collected from the signing of the informed consent form (ICF) until last AT follow up visit
Change in total score and domain scores | From Day 1 to Day 421; From Week -24 to Day -1
  Change in total score and domain scores is assessed by the Hemophilia Joint Health Score
Target joints resolution | At Day 421
  Target joints resolution assessed per ISTH criteria

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Investigational Site Number : 7920001, Istanbul
  - Investigational Site Number : 7920002, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC17905 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26981&tenant=MT_SNY_9011